CLINICAL TRIAL: NCT05932602
Title: The AVEIR DR Coverage With Evidence Development (DRIVE) Study
Brief Title: AVEIR DR Coverage With Evidence Development (CED) Study
Status: Recruiting | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: ABT-CIP-1020548
Record Dates: First submitted 2023-06-23; First posted 2023-07-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Cardiac Pacemaker; Arrythmia; Bradycardia
Keywords: dual chamber; sick sinus rhythm; pacemaker; AV Block
MeSH Terms: conditions — Arrhythmias, Cardiac; Bradycardia; Atrioventricular Block

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Aveir DR Leadless Pacemaker System: This study will utilize real-world data from patients implanted with the Aveir DR Leadless Pacemaker System. No device intervention is required in this study.
  Interventions: Device: Aveir DR Leadless Pacemaker System
- Dual Chamber Transvenous Pacemaker: This study will utilize real-world data from patients implanted with a dual-chamber transvenous pacemaker as a comparator to the Aveir DR LP system study arm. No device intervention is required in this study.
  Interventions: Device: Dual Chamber Transvenous Pacemaker

INTERVENTIONS:
Device: Aveir DR Leadless Pacemaker System — This study will utilize real-world data from patients implanted with the Aveir DR Leadless Pacemaker System. No device intervention is required in this study.
  Groups: Aveir DR Leadless Pacemaker System
Device: Dual Chamber Transvenous Pacemaker — This study will utilize real-world data from patients implanted with a dual-chamber transvenous pacemaker as a comparator to the Aveir DR LP system study arm. No device intervention is required in this study.
  Groups: Dual Chamber Transvenous Pacemaker

SUMMARY:
The purpose of this coverage with evidence development (CED) study is to evaluate complications and long-term health outcomes of the dual chamber Aveir Leadless Pacemaker device (aka Aveir™ DR LP system).

DETAILED DESCRIPTION:
This CED study utilizes a real-world evidence (RWE) method merging multiple real-world datasets from Abbott and the Center for Medicare Services to assess Aveir DR LP health outcomes among Medicare beneficiaries.

The study will enroll all Medicare patients with continuous claims data implanted with the Aveir DR LP system or a dual-chamber transvenous pacemaker system from any manufacturer.

Due to the RWE data collection methods used in this study, a central institutional review board (IRB) approved informed consent waiver has been granted. Due to this waiver and the sponsor's use of the central IRB, individual hospitals are not required to consent patients or complete local IRB submissions for this RWE study.

ELIGIBILITY:
Inclusion Criteria:

* Medicare beneficiaries implanted with an Aveir DR leadless pacemaker on or after the study start date (i.e., the date of Aveir DR market approval) will be included in the study.

OR

Medicare beneficiaries implanted with a full system (e.g. lead and generator) dual-chamber transvenous pacemaker on or after the study start date

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study cohort will include all Medicare patients with continuous claims data implanted with an Aveir DR leadless pacemaker or a full-system dual-chamber transvenous pacemaker (from any manufacturer) in any US location
Sampling Method: Non-Probability Sample
Enrollment: 2812 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Acute device related complication rate | 30 days
  Assess the acute (30-day) complication rate of the Aveir DR LP, compared to dual chamber transvenous pacemakers. An acute complication is defined as a peri-procedural, device-related adverse event occurring within 30 days post-implant.
Two-year survival rate | 2 years
  Assess (2-year) survival rate of subjects implanted with an Aveir DR LP, compared to dual chamber transvenous pacemakers.

SECONDARY OUTCOMES:
Chronic complication rate | 6 months
  Assess the chronic (6-month) complication rate of the Aveir DR LP, compared to dual chamber transvenous pacemakers. A chronic complication is defined as a post-procedural, device-related adverse event that requires invasive intervention to resolve, occurring more than 30 days through six months post implant.
Device-related re-intervention rates | 2 years
  Assess (2-year) device-related re-intervention rates of the Aveir DR LP, compared to dual chamber transvenous pacemakers

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Harbert, Study Director — Abbott
Locations (1):
- Abbott, Sylmar, California, United States